CLINICAL TRIAL: NCT01610856
Title: A Randomized Prospective Trial Comparing Single Dose Polyethylene Glycol-based Lavage Versus Split Dose Polyethylene Glycol-based Lavage in the Preparation of Patients Undergoing Colonoscopy
Brief Title: Single Dose Versus Split Dose Polyethylene Glycol-based Colonic Lavage for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Alaa Rostom, MD MSc FRCPC, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 21972; Ethics ID 21972 (Other: University of Calgary Ethics ID)
Record Dates: First submitted 2012-05-30; First posted 2012-06-04 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Colonoscopy Preparation
Keywords: bowel preparation; bowel purgative; bowel cleansing; colonoscopy
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEG - 4 L (Experimental): 4 Litres PEG bowel preparation given the day prior to colonoscopy with a clear fluid diet
  Interventions: Drug: Polyethylene Glycol
- Split Dose PEG (Active Comparator): 4 Litres of Colyte given as two split doses of 2L each either the day before colonoscopy 8 hours apart in the case of an AM colonoscopy or in the case of an afternoon colonoscopy given 5PM the day before and 6:00AM the day of the colonoscopy
  Interventions: Drug: polyethylene glycol

INTERVENTIONS:
Drug: Polyethylene Glycol — 4 Litres of polyethylene glycol bowel preparation solution
  Other Names: co-lyte; Go-lyte; PEG
  Arms: PEG - 4 L
Drug: polyethylene glycol — Polyethylene glycol 4L given in two split doses of 2L each
  Other Names: PEG; Co-lyte; Go-lyte
  Arms: Split Dose PEG

SUMMARY:
Proper bowel cleansing prior is an essential requirement for the conduct of colonoscopy. However, due to the nature of cleansing process, the ideal bowel cleansing preparation remains elusive.

The objective of this study is to compare the efficacy, safety and tolerability of oral polyethylene glycol lavage given either as a single dose or split dose. The study will be a randomized controlled single blind two group study. The primary study outcomes will be the previously validated Ottawa bowel preparation score.

DETAILED DESCRIPTION:
All patients between the age of 50 and 75 years referred to the Forzani & MacPhail Colorectal Cancer Screening Centre in Calgary, Alberta, Canada for colonoscopy will be considered for inclusion. During pre-assessments at the clinic, patients will be asked to participate in the study by a nurse clinician. If they agree - final consent will be obtained by a gastroenterologist along with consent for the colonoscopy. Those not interested in participating will simply receive their physicians standard bowel preparation protocol. There will be no coercion of any sort.

Patients with acute coronary syndrome, congestive heart failure, unstable angina, known or suspected renal failure, ascites, megacolon, known or suspected bowel obstruction, or other comorbidities that may prevent colonoscopy will be excluded. Patients will also be excluded if they previously had partial or subtotal colectomy or if the colonoscopy is warranted for the evaluation of diarrhea.

Enrollment of participants will be performed with block randomizations of 8 stratified by AM versus PM procedure time using a computer-generated table, with allocation concealment maintained through the use of consecutively numbered sealed envelopes. Colonoscopists and investigators will be blinded to allocation groups. Patients will be allocated to one of two groups: (1) 4L PEG day prior to procedure; (2) 4L of PEG split in two 2L doses

A study assistant will assign patients to their group and instruct them on the proper use of their assigned bowel preparation method. Patients will be given a tolerability questionnaire, that was modified from a previously reported questionnaire, to be completed once their bowel preparation is finished and before coming to the hospital for the colonoscopy. Patient concerns or questions regarding the preparation will be directed toward the assistant as opposed to their gastroenterologist, so as to avoid unblinding the gastroenterologist.

Outcomes

The previously validated Ottawa bowel preparation scale80 will be used to assess the quality of bowel cleanliness. Each of the right, mid and rectosigmoid colon is rated on a 5-point scale (0-4). In addition, a complete 3-point rating for overall colonic fluid is assessed resulting in an overall score range of 0 to 14. An excellent preparation with little fluid would score 0 to 1; a good preparation, 2 to 4; while scores higher than 4 would indicate progressively worsening bowel preparations. A completely unprepared colon would score 11 to 14, depending on the amount of colonic fluid.

Colonoscopy will be performed in a standard fashion and endoscopists will rate the bowel-preparation quality during the procedure and record the result on a separate standardized form.

Secondary outcomes will include a previously validated tolerability questionnaire and patient and investigator reported adverse events.

ELIGIBILITY:
Inclusion Criteria:

* All patients between the age of 50 and 75 years referred to the Forzani & MacPhail Colorectal Cancer Screening Centre in Calgary, Alberta, Canada for colonoscopy will be considered for inclusion.

Exclusion Criteria:

* patients with acute coronary syndrome,
* congestive heart failure,
* unstable angina,
* known or suspected renal failure,
* ascites,
* megacolon,
* known or suspected bowel obstruction, or
* other comorbidities that may prevent colonoscopy will be excluded. Patients will also be excluded if they previously had partial or subtotal colectomy or if the colonoscopy is warranted for the evaluation of diarrhea.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The Ottawa Bowel Preparation Score | Measured at time of Colonoscopy
  A validated scale. Each of the right, mid and rectosigmoid colon is rated on a 5-point scale (0-4). In addition, a complete 3-point rating for overall colonic fluid is assessed resulting in an overall score range of 0 to 14. An excellent preparation with little fluid would score 0 to 1; a good preparation, 2 to 4; while scores higher than 4 would indicate progressively worsening bowel preparations. A completely unprepared colon would score 11 to 14, depending on the amount of colonic fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Rostom, MD MSc FRCPC, Principal Investigator — University of Calgary
Locations (1):
- Forzani & MacPhail Colon Cancer Screening Centre, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Mohamed R, Hilsden RJ, Dube C, Rostom A. Split-Dose Polyethylene Glycol Is Superior to Single Dose for Colonoscopy Preparation: Results of a Randomized Controlled Trial. Can J Gastroenterol Hepatol. 2016;2016:3181459. doi: 10.1155/2016/3181459. Epub 2016 Apr 13. PMID 27446836